CLINICAL TRIAL: NCT06258343
Title: Examination of Intact and Amputated Extremity Thermographic Values in Individuals With Transtibial Amputation
Brief Title: Extremity Thermographic Values in Individuals With Transtibial Amputation
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Collaborators: Gulhane School of Medicine (Other); Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Senay Cerezci Duygu, Asst. Prof., Baskent University
Other Study IDs: 2022-1274
Record Dates: First submitted 2024-01-28; First posted 2024-02-14 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2024-08

CONDITIONS: Amputees; Amputation; Amputation Stump; Amputation of Knee; Vascularisation
MeSH Terms: conditions — Neovascularization, Pathologic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to compare thermographic values in the knee region of the healthy extremity and the amputated extremity and learn about the relationship between thermographic value and pain in the knee region of the amputated extremity. The main questions it aims to answer are:

1. Do thermal values in the knee region of the amputated extremity and the intact extremity differ in individuals with transtibial amputation?
2. Is there a relationship between the pain felt in the knee region of the amputated limb and the difference in thermal values between the extremities in individuals with transtibial amputation?

DETAILED DESCRIPTION:
With amputation, anatomical and vascular changes occur in the distal part of the remaining limb. At this point, for individuals with amputation at the transtibial level, the knee joint in the amputated extremity is of critical importance as it is the most distal joint. While there is evidence that thermal changes observed in the knee region may be related to possible degeneration or pathological processes, there is not enough research on the amputee population. Considering that individuals who have undergone lower extremity amputation are at greater risk than the general population for many health problems and considering the current evidence, we think that the evaluation of skin temperature, which is an indicator of cutaneous circulation, may be an important indicator in taking precautions for degenerative knee diseases. With the planned study, lower extremity temperature profiles and their relationship with knee pain will be evaluated for the first time during the post-amputation period. Thermal infrared non-contact thermometer, which is non-invasive, cheap and easy to apply, will be used for the first time in lower extremity temperature measurements of amputees.

Objectives of the study,

* Thermal analysis results of both extremities will be compared and it will be investigated whether there is a difference between thermal values, which is one of the indicators of cutaneous blood flow;
* By comparing the thermal values, it will be determined whether the thermal values differ in the amputee limb that has undergone major trauma and is exposed to prosthetic material that applies continuous compression,
* The relationship between nociceptive pain and phantom pain felt in the knee region of the amputated limb and the thermal value difference between the extremities will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Having a unilateral below knee level amputation,
* Using a prosthesis and being able to walk with the prosthesis,
* Not having undergone any surgery related to the knees.

Exclusion Criteria:

* Having bilateral amputation,
* Not being able to walk 10 minutes independently,
* Failure to consent to measurement of knee thermal temperature.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with unilateral transitibial amputation
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Skin Temperature | 30 minutes
  In both knees, 3 measurements will be taken at the center of the patella, the tibialis anterior muscle trunk (10 cm distal to the tibial tubercle and 2 cm lateral to the anterior border of the tibia) and distal to the limb. Room temperature will be recorded simultaneously. Measurements will be recorded in Celsius. The study will follow the recently published 15-point TISEM consensus statement on the measurement of human Tsk. Within the scope of the study, temperature measurements will be performed using a Medisana 48620 Infrared Non-Contact Thermometer (MEDISANA, FTN, Hilden, Germany).

SECONDARY OUTCOMES:
Knee Pain | 10 minutes
  The presence of pain in both knees, pain intensity and localization of pain will be questioned. To determine the presence of pain sensation in the knee region of the patients, the presence or absence of pain sensation in the knee of the intact and amputated extremity will be questioned. In the presence of pain sensation, the 'Visual Analog Scale' will be used to assess the severity of pain in the intact knee and the amputated knee.
  For pain intensity assessment with the Visual Analog Scale, a 10 cm long line is drawn. The starting and ending points of the line are numbered 0 and 10. Individuals are asked to mark the intensity of the pain they feel on the scale, indicating that a value of 0 indicates absence of pain and a value of 10 indicates unbearable severe pain. The area marked by the individuals is then measured with a ruler and recorded as pain intensity.
Phantom Sensation and Phantom Pain | 20 minutes
  The presence of phantom limb sensation will be questioned. If there is phantom limb sensation, individuals will be asked to describe their phantom limb sensation with open-ended questions and to provide information about the position of their limbs (fixed or mobile, in anatomical position or in anatomically impossible position), and whether they feel shortening/shrinking or any other condition in their limbs and the presence of telescope phenomenon will be questioned.
  The presence or absence of phantom pain will be questioned. If phantom pain is experienced, individuals will be asked to provide information about the area of pain, the frequency/type of pain and to complete the "Short Form Mc-Gill Pain Scale (SF-MPQ)". The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Senay Cerezci Duygu, Ankara, Keçiören, Turkey (Türkiye)